CLINICAL TRIAL: NCT01274052
Title: Reduced Postprandial GLP-1 Response in Gestational Diabetes Mellitus: a Fully Reversible Phenomenon
Brief Title: Study of Postprandial Incretin Response in Women With Gestational Diabetes
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: The Danish Diabetes Association (Other); Aase and Ejnar Danielsens Foundation (Other); The Novo Nordic Foundation (Other)
Responsible Party: Filip K. Knop, MD PhD, Department of Internal Medicine F, University Hospital, Gentofte, Copenhagen
Other Study IDs: KA-060015
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Gestational diabetes mellitus; Meal test; Incretin hormones; Glucagon-like peptide-1 (GLP-1); Glucose-dependent insulinotropic polypeptide; Insulin; C-peptide; Glucagon
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gestational Diabetes Mellitus: Women with Gestational Diabetes Mellitus
  Interventions: Other: Meal test
- Normal Glucose Tolerance: Women with Normal Glucose Tolerance
  Interventions: Other: Meal test

INTERVENTIONS:
Other: Meal test — Liquid meal test

SUMMARY:
The researchers investigated nineteen pregnant women in third trimester and again postpartum. At the experimental days we performed a mealtest and drew blood for analyses of glucagon-like peptide-1 (GLP-1), glucose-dependent insulinotropic polypeptide (GIP), insulin, C-peptide and glucagon.

The researchers aimed to investigate whether women with gestational diabetes mellitus exhibit decreased postprandial GLP-1 responses, and if so, whether this deficiency ceases following delivery when normal glucose tolerance is reestablished.

DETAILED DESCRIPTION:
The researchers investigated nineteen pregnant women in third trimester and again postpartum. At the experimental days we performed a mealtest and drew blood for analyses of glucagon-like peptide-1 (GLP-1), glucose-dependent insulinotropic polypeptide (GIP), insulin, C-peptide and glucagon.

The researchers aimed to investigate whether women with gestational diabetes mellitus exhibit decreased postprandial GLP-1 responses, and if so, whether this deficiency ceases following delivery when normal glucose tolerance is reestablished.

ELIGIBILITY:
Inclusion Criteria:

* Normal haemoblobin
* Willingness to participate

Exclusion Criteria:

* First degree relative with diabetes
* Diabetes before pregnancy
* Positive islet cell- and GAD-65 autoantibodies

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Healthy pregnant woman were examined with a 75 g oral glucose tolerance test. Subjects with plasma glucose (PG) values at 120 min >9.0 mmol/l were diagnosed with gestational diabetes and subjects with PG <9.0 mmol/l were enrolled as healthy controls.
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2007-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD PhD, Principal Investigator — Diabetes Research Division, Gentofte Hopsital
Locations (1):
- Department of Internal Medicine, Glostrup Hospital, Glostrup Municipality, Denmark

REFERENCES:
- [Derived] Hare KJ, Bonde L, Svare JA, Randeva HS, Asmar M, Larsen S, Vilsboll T, Knop FK. Decreased plasma chemerin levels in women with gestational diabetes mellitus. Diabet Med. 2014 Aug;31(8):936-40. doi: 10.1111/dme.12436. Epub 2014 Apr 1. PMID 24628007